CLINICAL TRIAL: NCT05468996
Title: Median Effective Dose of Remimazolam for Sedation in Elderly Patients Undergoing Lower Limb Surgery Under Spinal Anesthesia
Brief Title: Median Effective Dose of Remimazolam for Sedation in Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Won Uk, Koh, Associate Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-1869
Record Dates: First submitted 2022-05-12; First posted 2022-07-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Sedative
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- young-old group (Active Comparator): a group of patients who are 60 to 74 years old
  Interventions: Drug: Remimazolam
- old-old group (Active Comparator): a group of patients who are equal or older than 75 years
  Interventions: Drug: Remimazolam
- young adult group (Active Comparator): a group of patients who are 20-59 years old
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — A loading dose of remimazolam is 1mg/kg/hr. When sedation is achieved, the dose of remimazolam is adjusted to the assigned dose. The maintenance dose of remimazolam begins at 1.0mg/kg/hr. When the maintenance is not successful during the surgery, the maintenance dose will be increased by 0.1-0.2mg/kg/hr in the next patient. When the maintenance is successful, the dose will be decreased by 0.1-0.2mg/kg/hr. (maximal dose: 2mg/kg/hr)

SUMMARY:
Currently used drugs for monitored general anesthesia include propofol, midazolam, and dexmedetomidine. Each drug has different advantages and disadvantages. Remimazolam causes a relatively small decrease in blood pressure, and it has no injection pain. In addition, remimazolam has a very short onset time, and even after the continuous infusion, the onset of remimazolam is fast, and even after continuous injection, the effect disappeared very quickly due to the short context-sensitive half time. And through continuous infusion, the patient's depth of anesthesia can be maintained constant. In addition, the short duration of action and the ability to quickly reverse the effect of flumazenil suggest that remimazolam can be used effectively under general anesthesia as well as under general anesthesia. Remimazolam can be used as a continuous infusion for general anesthesia. However, it has also been reported to be used for sedation by continuous infusion or divided intravenous infusion. However, the effective maintenance dose of remimazolam for sedation without mechanical ventilation has not been established. In addition, age might be an important factor for determining the appropriate dose of remimazolam.

In this study, we aim to identify the median effective dose of remimazolam for maintaining sedation in elderly patients undergoing lower limb surgery under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age: equal or older than 20 years
* ASA PS: 1-3
* patients who are scheduled to undergo lower limb surgery under spinal anesthesia with sedation using remimazolam

Exclusion Criteria:

* Patients who refuse to participate in this study
* Patients with hypersensitivity to benzodiazepine or flumazenil
* Patients with severe renal/hepatic disease
* Patients with drug/alcohol abuse
* Patients who take antidepressants, anticonvulsants, psychoactive drugs chronically
* Patients with difficulty in communication
* Patients with severe obstructive sleep apnea or other airway problems
* Patients contraindicated to regional anesthesia
* Patients judged to be inappropriate for this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
success or failure of sedation maintenance | throughout the surgery
  MOAA/S score of 3 or less (MOAA/S: Modified Observer's Alertness/Sedation scale) Awake (5) - Unresponsive (0)

SECONDARY OUTCOMES:
respiratory depression | throughout the surgery
  respiratory rate equal or less than 6 time per minute

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea